CLINICAL TRIAL: NCT02463227
Title: A Phase I, Open-Label Study of the Safety, Pharmacokinetics, and Antiviral Activity of a Human Monoclonal Antibody, VRC-HIVMAB060-00-AB (VRC01), With Broad HIV-1 Neutralizing Activity, Administered Intravenously to HIV-Infected Adults Undergoing a Brief Analytical Treatment Interruption
Brief Title: Evaluating the Safety, Pharmacokinetics, and Antiviral Activity of a Human Monoclonal Antibody (VRC01) in HIV-Infected Adults Undergoing a Brief Treatment Interruption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5340; 11998 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2015-05-29; First posted 2015-06-04 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2017-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — VRC01 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VRC01 (Experimental): Participants received an IV infusion of 40 mg/kg of VRC01 on study days 0, 21, and 42.
  Interventions: Biological: VRC01

INTERVENTIONS:
Biological: VRC01 — 40 mg/kg of VRC01 administered IV in 100 mL of 0.9% sodium chloride for injection, USP.
  Administered over about 30 to 60 minutes using a volumetric pump.
  Other Names: VRC-HIVMAB060-00-AB

SUMMARY:
The purpose of this study was to evaluate the safety, tolerability, pharmacokinetics (PK), and antiviral activity of an antibody (called VRC01) in HIV-infected adults whose HIV was well-controlled with HIV medicines. The study examined whether VRC01 controlled or delayed the return of HIV viremia when the participants' HIV medicines were briefly stopped during the study.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the safety, tolerability, pharmacokinetics (PK), and antiviral activity of a human monoclonal antibody, VRC-HIVMAB060-00-AB (known as VRC01), in HIV-infected adults whose HIV was well-controlled with antiretroviral therapy (ART). The study examined whether VRC01 delayed or prevented the return of HIV viremia in participants who underwent a brief analytical treatment interruption (ATI).

The study enrolled HIV-infected participants 18 years and older who were on ART (ART was not provided by the study). At a pre-entry study visit, participants underwent blood collection, a leukapheresis procedure, and a rectal biopsy. The study lasted about 34 weeks and proceeded in three stages: Step 1 (approximately 9 weeks), Step 2 (approximately 12 weeks), and Step 3 (approximately 13 weeks).

During Step 1, participants received three doses of VRC01 via intravenous (IV) infusion. The first dose of VRC01 was given on day 0. Seven days after receiving this first dose of VRC01, participants discontinued ART. Participants received the second and third doses of VRC01 at days 21 and 42, respectively. For 7 days after each VRC01 IV infusion, participants monitored and recorded their temperature and any symptoms. In addition to the 3 infusion study visits, participants attended weekly visits from day 7 through approximately day 63 (week 9).

Participants entered Step 2 of the study and resumed ART when they had a confirmed CD4+ T-cell count of less than 350 cells/μL or a confirmed return of HIV-1 viremia, defined per protocol as an HIV-1 RNA measurement of greater than or equal to 200 copies/mL followed by a confirmatory measurement of greater than or equal to 1000 copies/mL or three consecutive HIV-1 RNA measurements of over 200 copies/mL.

Step 2 study visits occurred on the day ART was resumed (Step 2, entry) and every four weeks thereafter (approximately at Step 2, weeks 4, 8, and 12) until a participant's HIV viral load decreased to less than 50 copies/mL.

Throughout the study, visits included clinical assessments and blood collection. Some blood was stored for future testing. Some study visits included the collection of oral, rectal, and (for women) cervical secretion samples. On day 63, participants underwent another leukapheresis procedure and a rectal biopsy.

Participants who completed Step 2 may have optionally entered Step 3 for additional testing. Entry into Step 3 occurred at least 3 months after the participant had completed Step 2. Step 3 participants had additional study visits for a leukapheresis procedure, a rectal biopsy, and clinical follow up.

ELIGIBILITY:
Step 1 Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load (VL). More information on this criterion can be found in the protocol.
* Ability and willingness of participant or legal representative to provide informed consent
* Clinically stable on their first or second ART regimen that includes a boosted protease inhibitor or an integrase inhibitor. The current regimen should have been stable for 8 weeks at the time of entry. Changes while the patient HIV viral load was undetectable did not count toward the number of ART regimens used, (for example, an individual switching from a non-nucleoside reverse transcriptase inhibitor (NNRTI)-based regimen to an integrase inhibitor based regimen while the HIV viral load is undetectable would still be on their first regimen).
* HIV-1 RNA that is less than 50 copies/mL using a Food and Drug Administration (FDA)-approved assay performed by any laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent within 45 days prior to study entry
* HIV-1 RNA less than 50 copies/mL using a FDA-approved assay for at least 24 weeks prior to study entry performed by any laboratory that had a CLIA certification or its equivalent. More information on this criterion can be found in the protocol.
* Screening CD4+ T-cell count greater than or equal to 450 cells/μL within 45 days prior to study entry
* Nadir CD4+ T-cell count greater than 200 cells/μL
* Willingness to have blood samples collected, stored indefinitely, and used for study-related research purposes
* The following laboratory values obtained within 45 days prior to enrollment:

  * Absolute neutrophil count (ANC) greater than or equal to 1000 cells/mm^3
  * Hemoglobin greater than or equal to 12.0 g/dL for men and greater than or equal to 11.0 g/dL for women
  * Platelet count greater than or equal to 100,000/mm^3
  * Creatinine clearance greater than or equal to 60 mL/min estimated by the Cockcroft-Gault equation. More information on this criterion can be found in the protocol.
  * Alanine aminotransferase (ALT) less than or equal to 2.0 times the upper limit of normal (ULN)
* At least eight participants had availability of plasma or serum specimen before the initiation of ART either in the Center for AIDS Research (CFAR) repository of the University of Pennsylvania, University of Alabama, or in the AIDS Clinical Trials Group (ACTG) central repository
* For females of reproductive potential (i.e., women who have not been post-menopausal for at least 24 consecutive months; who had menses within the preceding 24 months; or women who had not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy), negative urine pregnancy test (with a sensitivity of 15 to 25 mIU/mL) within 48 hours prior to screening and entry. More information on this criterion can be found in the protocol.
* Contraceptive methods were required for female participants of reproductive potential. Female participants of reproductive potential and their male partners MUST HAVE appropriately used at least two contraceptives, with one method being highly effective and the other method being either highly effective or less effective. More information on this criterion, including a list of acceptable contraceptive options, can be found in the protocol.
* Contraceptive methods were required for female partners of reproductive potential of male study participants on study drug. Female partners of reproductive potential of male study participants and/or their male partners MUST HAVE appropriately used at least two contraceptives, with one method being highly effective and the other method being either highly effective or less effective. More information on this criterion, including a list of acceptable contraceptive options, can be found in the protocol.
* Negative hepatitis B surface antigen (HBsAg) result obtained within 6 months prior to study entry
* Hepatitis C virus (HCV) antibody negative result within 6 months prior to entry, or if the HCV antibody result was positive, a negative HCV RNA obtained within 6 months prior to study entry
* Adequate venous access in at least one arm

Step 2 Inclusion Criteria:

* Entry into Step 1 of this study (A5340)
* Receipt of at least one dose or partial dose of VRC01 in Step 1
* Reinitiating ART for protocol or non-protocol-defined reasons. More information on this criterion can be found in the protocol.

Step 3 Inclusion Criteria:

* Entry into and completion of Step 2 of this study (A5340) at least 3 months prior
* HIV-1 RNA less than 50 copies/ml at pre-entry visit
* Ability and willingness of participant or legal representative to provide informed consent
* Willingness to have blood samples/specimens collected, stored indefinitely, and used for study-related research purposes
* Adequate venous access in at least one arm

Step 1 Exclusion Criteria:

* Previous receipt of humanized or human monoclonal antibody whether licensed or investigational
* Weight greater than 115 kg or less than 53 kg
* History of an AIDS-defining illness
* Ongoing AIDS-related opportunistic infection (including oral thrush)
* History of a severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis in the 2 years prior to enrollment
* Currently breastfeeding
* Receipt of other investigational study agent within 30 days prior to enrollment
* Treatment with systemic glucocorticoids (e.g., prednisone or other glucocorticoid) or other immunomodulators (other than nonsteroidal anti-inflammatory drugs [NSAIDs]) within 30 days prior to enrollment
* Any other chronic or clinically significant medical condition that in the opinion of investigator would have jeopardized the safety or rights of the participant, including, but not limited to diabetes mellitus type I, OR clinically significant forms of drug or alcohol abuse, severe asthma, autoimmune disease, uncontrolled hypertension, liver disease, psychiatric disorders, heart disease, or cancer
* Treatment during acute infection (i.e., treatment within 6 months of acute infection)
* Current use of a NNRTI

Step 2 Exclusion Criteria:

* Non-participation in Step 1

Step 3 Exclusion Criterion:

* Non-participation in Step 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Study Chair — University of Pennsylvania
Locations (2):
- United States (2):
  - Alabama CRS, Birmingham, Alabama
  - Penn Therapeutics, CRS, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Zhou T, Georgiev I, Wu X, Yang ZY, Dai K, Finzi A, Kwon YD, Scheid JF, Shi W, Xu L, Yang Y, Zhu J, Nussenzweig MC, Sodroski J, Shapiro L, Nabel GJ, Mascola JR, Kwong PD. Structural basis for broad and potent neutralization of HIV-1 by antibody VRC01. Science. 2010 Aug 13;329(5993):811-7. doi: 10.1126/science.1192819. Epub 2010 Jul 8. PMID 20616231
- [Background] Li Y, O'Dell S, Walker LM, Wu X, Guenaga J, Feng Y, Schmidt SD, McKee K, Louder MK, Ledgerwood JE, Graham BS, Haynes BF, Burton DR, Wyatt RT, Mascola JR. Mechanism of neutralization by the broadly neutralizing HIV-1 monoclonal antibody VRC01. J Virol. 2011 Sep;85(17):8954-67. doi: 10.1128/JVI.00754-11. Epub 2011 Jun 29. PMID 21715490
- [Background] U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS. Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0. [November 2014]. Available from: http://rsc.tech-res.com/docs/default-source/safety/daids_ae_grading_table_v2_nov2014.pdf
- [Background] Manual for Expedited Reporting of Adverse Events to DAIDS, Version 2.0, January 2010.
- [Result] Bar KJ, Sneller MC, Harrison LJ, Justement JS, Overton ET, Petrone ME, Salantes DB, Seamon CA, Scheinfeld B, Kwan RW, Learn GH, Proschan MA, Kreider EF, Blazkova J, Bardsley M, Refsland EW, Messer M, Clarridge KE, Tustin NB, Madden PJ, Oden K, O'Dell SJ, Jarocki B, Shiakolas AR, Tressler RL, Doria-Rose NA, Bailer RT, Ledgerwood JE, Capparelli EV, Lynch RM, Graham BS, Moir S, Koup RA, Mascola JR, Hoxie JA, Fauci AS, Tebas P, Chun TW. Effect of HIV Antibody VRC01 on Viral Rebound after Treatment Interruption. N Engl J Med. 2016 Nov 24;375(21):2037-2050. doi: 10.1056/NEJMoa1608243. Epub 2016 Nov 9. PMID 27959728
- [Derived] Weir IR, Harrison LJ. An evaluation of confidence intervals for a cumulative proportion to enable decisions at interim reviews of single-arm trials. Contemp Clin Trials. 2024 Mar;138:107453. doi: 10.1016/j.cct.2024.107453. Epub 2024 Jan 20. PMID 38253253
- [Derived] Salantes DB, Zheng Y, Mampe F, Srivastava T, Beg S, Lai J, Li JZ, Tressler RL, Koup RA, Hoxie J, Abdel-Mohsen M, Sherrill-Mix S, McCormick K, Overton ET, Bushman FD, Learn GH, Siliciano RF, Siliciano JM, Tebas P, Bar KJ. HIV-1 latent reservoir size and diversity are stable following brief treatment interruption. J Clin Invest. 2018 Jul 2;128(7):3102-3115. doi: 10.1172/JCI120194. Epub 2018 Jun 18. PMID 29911997

RESULTS

PARTICIPANT FLOW:
Groups:
- VRC01: Participants received an IV infusion of 40 mg/kg of VRC01 on study days 0, 21, and 42.
  VRC01: 40 mg/kg of VRC01 administered IV in 100 mL of 0.9% sodium chloride for injection, USP.
  Administered over about 30 to 60 minutes using a volumetric pump.
Period: Overall Study
Arm/Group | VRC01
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled.
Arm/Group | VRC01
Number analyzed (Participants) | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [34 to 44]
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 1
  30-39 years | 6
  40-49 years | 6
  50+ years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 6
  Black Non-Hispanic | 6
  Hispanic (Regardless of Race) | 2
Region of Enrollment [Number; unit: participants]
  United States | 14
Intravenous Drug History [Count of Participants; unit: Participants]
  Never | 13
  Previously | 1
Weight [Median (Inter-Quartile Range); unit: kilograms] | 86 [77 to 102]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 28.3 [25.4 to 31.3]
HIV-1 RNA [Count of Participants; unit: Participants] — The categories < 20 copies/mL and < 40 copies/mL are mutually exclusive. These categories represent results below the limit of detection from different assays used to assess HIV-1 RNA.
  Participants
    < 20 copies/mL | 10
    < 40 copies/mL | 2
    = 40 copies/mL | 1
    = 50600 copies/mL | 1
CD4 Cell Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 896 [579 to 1053]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced a Grade 3 or Higher Systemic (i.e., Not a Local Reaction) Adverse Event (AE) That is Possibly, Probably, or Definitely Related to the Administration of the VRC01 Antibody
Description: The primary safety outcome examined the occurrence of a Grade 3 or higher systemic (i.e., not a local reaction) adverse event (AE) possibly, probably, or definitely related to the administration of the VRC01 antibody. The DAIDS AE Grading Table (V2.0) was used.
Time Frame: Measured from entry through week 21 (Steps 1 and 2)
Population: All participants exposed to study treatment (VRC01) were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VRC01
Number analyzed (Participants) | 14
percentage of participants | 0 [0 to 23]

2. Primary Outcome: Percentage of Participants Who Had a Confirmed HIV-1 RNA Greater Than or Equal to 200 Copies/mL at Week 8 of the Analytical Treatment Interruption (ATI) or Indication to Re-initiate ART Prior to Week 8 of the ATI
Description: The primary efficacy outcome is the percentage of participants who had a confirmed HIV-1 RNA greater than or equal to 200 copies/mL at week 8 of the analytical treatment interruption (ATI) or indication to re-initiate ART prior to week 8 of the ATI.
Time Frame: Measured at Weeks 1, 2, 3, 4, 5, 6, 7, and 8 of the ATI
Population: Per protocol, the analysis population was limited to participants who received all scheduled VRC01 infusions and underwent an ATI according to protocol.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | VRC01
Number analyzed (Participants) | 13
percentage of participants | 92 [68 to 99.6]

3. Secondary Outcome: Measured Value of Plasma VRC01 at the Time of Rebound
Description: Measured value of plasma VRC01, measured in micrograms per milliliter, at the time of rebound. Rebound is defined as the point in time when plasma HIV-1 RNA surpassed 40 copies/mL.
Time Frame: Measured from entry through week 21 (Steps 1 and 2)
Population: as for outcome 2
Measure: Median (Full Range); unit: micrograms/mL
Arm/Group | VRC01
Number analyzed (Participants) | 13
micrograms/mL | 127 [25 to 255]

4. Secondary Outcome: Measured Values of VRC01 in Plasma in the First 8 Weeks of the Analytical Treatment Interruption (ATI)
Description: Measured values of plasma VRC01, measured in micrograms per milliliter, through week 8 of the ATI. The median and range of all VRC01 measurements taken in the first 8 weeks of the ATI were reported.
Time Frame: Measured at weeks 1, 2, 3, 4, 5, 6, 7, and 8 of the ATI
Population: as for outcome 2
Measure: Median (Full Range); unit: micrograms/mL
Arm/Group | VRC01
Number analyzed (Participants) | 13
micrograms/mL | 175 [68 to 1494]

5. Secondary Outcome: Percentage of Participants Who Had a Confirmed HIV-1 RNA Greater Than or Equal to 200 Copies/mL at Week 4 of the ATI or Indication to Reinitiate ART Prior to Week 4 of the ATI
Description: The secondary efficacy outcome was the percentage of participants who had a confirmed HIV-1 RNA greater than or equal to 200 copies/mL at week 4 of the ATI or indication to reinitiate ART prior to week 4 of the ATI.
Time Frame: Measured at weeks 1, 2, 3, and 4 of the ATI
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | VRC01
Number analyzed (Participants) | 13
percentage of participants | 62 [35 to 83]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from entry throughout the study, up to week 34.
Description: The protocol required reporting of laboratory results and signs/symptoms grade ≥ 2, grade < 2 solicited signs/symptoms from the infusion report card, laboratory results and signs/symptoms that led to a change in VRC01 infusion, and diagnoses identified by the ACTG criteria for clinical events and other diseases since the last visit. The DAIDS AE Grading Table (V2.0) and Expedited AE Manual (V2.0) were used.
Arm/Group | VRC01
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 7/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VRC01 (N=14)
Pruritus (Skin and subcutaneous tissue disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Cervical radiculopathy (Nervous system disorders) | 1
Blood phosphorus abnormal (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood creatinine abnormal (Investigations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Onychomycosis (Infections and infestations) | 1
Infusion site induration (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No